CLINICAL TRIAL: NCT02109614
Title: A Pilot,Randomized Controlled-trial of Lipoprotein(a) Lowering for the Prevention of Aortic Valve Disease-translating Genomic Knowledge for Cardiovascular Prevention
Brief Title: Early Aortic Valve Lipoprotein(a) Lowering Trial
Acronym: EAVaLL
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: George Thanassoulis (Other)
Collaborators: Jewish General Hospital (Other); Laval University (Other); Quebec Heart Institute (Other)
Responsible Party: Sponsor-Investigator, George Thanassoulis, MD MSc FRCPC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: A00-M105-13A
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Aortic Stenosis and Lipoprotein(a) Levels
Keywords: lipoprotein(a); aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended release Niacin (Experimental): Taking 1500-2000mg niacin daily
  Interventions: Drug: Extended release Niacin
- No Naicin (Placebo Comparator): Placebo Comparator arm will be taking 1500mg of placebo daily
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Extended release Niacin — Arm will be taking 1500-2000mg of niacin daily to see if lipoprotein(a) levels are lowered and aortic stenosis does not increase.
  Arms: Extended release Niacin
Drug: Placebo Comparator — Placebo Comparator arm will be taking 1500mg of the placebo daily
  Arms: No Naicin

SUMMARY:
Aortic valve disease is the most common form of heart valve disease and is a major burden to society. Aortic valve disease is also expected to become more prevalent with the aging of the Canadian population. Currently, over 1 million individuals in North America have aortic stenosis, which is a narrowing of the aortic valve, and leads to symptoms of heart failure and sometimes death. Valve replacement with its potential costs and complications remains the only avenue for treatment, once symptoms develop. Despite the major importance of this disease, there are currently no medical treatments to prevent the development of aortic stenosis.The lack of preventative treatments stems in large part to a poor understanding of the causes of this disease.

Using cutting-edge genetic technologies, the investigators have recently identified that individuals with a genetic predisposition to elevations in a type of cholesterol not normally screened, called lipoprotein(a), have a much higher risk of developing aortic valve disease. The investigators have also shown that lipoprotein(a) causes hardening of the valve, a very early sign of valve narrowing. The investigators plan to evaluate in a randomized controlled trial whether lowering this unusual form of cholesterol at an early stage of this disease could slow or stop the development of aortic valve narrowing

The investigators are currently proposing a pilot project to evaluate the feasibility of this type of study. If successful, our proposed treatment would be notable in two ways. First, it would represent the first medical treatment to prevent valve disease, which could lead to major reductions in the societal burden of this important disease. And second, it would herald a major success for genomic medicine as it would represent one of the first treatments borne from recent genetic studies. In these ways, our proposal could significantly impact the health of many Canadians while also highlighting the innovative research performed in Canada.

Recruitment (n=238) for this project will be from the echocardiography laboratories of McGill University affiliated hospitals. Individuals with aortic sclerosis or mild aortic stenosis (aortic valve area [AVA] >1.5 cm2, mean gradient [MG] < 25 mmHG) and high Lp(a) will be eligible for inclusion into this proposed study.

DETAILED DESCRIPTION:
Screening: Potentially eligible participants from the echocardiography laboratory will be screened by a member of the research team for inclusion and exclusion criteria and will be asked to review and sign a consent form that explains the study.

Run-in: Participants with elevated Lp(a) and normal liver and renal indices, that meet all other inclusion and exclusion criteria will be started on low dose niacin (500 mg/d) for a 6 week run-in phase prior to randomization to assess tolerability and compliance to the intervention. The niacin dose will be increased by 500 mg increments weekly, as tolerated, to a maximum of 1500 mg/day (Participants who remain compliant >85% (by pill count and self-report) and who tolerate at least 1500 mg/d of niacin for at least 2 weeks will then undergo randomization to 1500 mg/d of immediate release niacin or matching placebo.

Randomization: will be performed via an Internet website where each participant will be given a unique identifier that matches the allocated drug kit.Blocking using random blocks of 2 and 4 will ensure that similar numbers of patients are randomized to the two arms of the study at each of the study centers.

The study will be double blind - neither patients, physicians, nor study personnel will know which participants are receiving active treatment.

After a 6-week run-in phase, participants able to tolerate the intervention will be randomized 1:1 to niacin extended release or placebo. After randomization, the treatment phase will be for 2 years (104 weeks). Data will be collected during 5 visits: (i) Randomization visit; (ii) 6-month follow-up visit; (iii) 12-month follow-up visit; (iv) 18-month follow-up visit; (v)Final visit (24-month).

(i) Randomization visit (baseline)

(1) Data Collected: A. Clinical and Biochemical Data B. Echocardiogram C. Blood Collection D. Cardiac CT

(ii) Follow-up visits (at 6, 12 and 18 months from randomization) Collection of clinical data (re: side-effects), compliance to therapy and blood.

(iii) Final visit (24 months) At the final visit, all usual data collected during the above follow-up visits will be obtained (including compliance, side-effects, etc). An echocardiogram, cardiac CT and a final blood test will also be obtained

1. Primary Endpoints

   a) Relative reduction in rates of calcium score progression by cardiac CT in individuals randomized to niacin as compared to those randomized to placebo.
2. Secondary Endpoints

   1. Number needed to screen to identify eligible participants
   2. Difference in mean change in Lp(a) levels between treatment arms
   3. Rates of progression in each arm by echocardiography at 1 and 2 years (Change in peak velocity (in m/s); Change in mean gradient (in mm Hg); Change in AVA (in cm2)
3. Tertiary Endpoints

   1. Compliance (as a proportion of pills taken/pills prescribed) with niacin treatment
   2. Rates of side-effects and other adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age >50 years and < 85 years
2. Aortic sclerosis OR mild AS

   * Aortic sclerosis: diffuse of focal (at least 2 areas) thickening or calcification (highly echodense lesions) on aortic leaflets seen in at least 2 contiguous views with normal leaflet excursion and peak aortic jet velocity < 2 m/s.
   * Mild AS: peak aortic jet velocity 2-3 cm/s, AVA >1.5cm2, mean gradient <25 m

     * Elevated Lp(a) > 50 mg/dL (>80th percentile).

Exclusion Criteria:

1. Current use or documented indication for niacin therapy or known niacin allergy/intolerance
2. Bicuspid valve, unicuspid valve or other congenital cardiac anomaly (except patent foramen ovale)
3. Known renal disease or more than mild renal dysfunction (Creatinine > 150 mmol/L or Creatinine clearance < 60).
4. Major comorbidities limiting life expectancy to < 2 years
5. Unable or unwilling to complete follow-up visits to 2 year
6. Diagnosed hepatic failure, cirrhosis, hepatitis or history of hepatic impairment (AST or ALT levels ³ 2 times upper limit of normal)
7. Newly diagnosed (< 2 months) or poorly controlled diabetes
8. Gout or use of anti-hyperuricemic medications

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Calcium score progression by cardiac CT in individuals randomized to niacin as compared to those randomized to placebo | 2 years

SECONDARY OUTCOMES:
Mean change in Lp(a) levels between treatment arms | 2 years

OTHER OUTCOMES:
Rates of valve disease progression by echocardiography at 1 and 2 years | 1 and 2 years
  Change in peak velocity (in m/s); Change in mean gradient (in mm Hg); Change in AV area (in cm2)
Drug compliance | At 6, 12, 18 and 24 months
  Pill count and drug diary
Side effects and adverse events | at 6, 12, 18 and 24 months
  all common and rare serious side-effects/adverse events will be monitored

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - MUHC - Montreal General Hospital, Montreal, Quebec
  - MUHC - Royal Victoria Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Thanassoulis G, Campbell CY, Owens DS, Smith JG, Smith AV, Peloso GM, Kerr KF, Pechlivanis S, Budoff MJ, Harris TB, Malhotra R, O'Brien KD, Kamstrup PR, Nordestgaard BG, Tybjaerg-Hansen A, Allison MA, Aspelund T, Criqui MH, Heckbert SR, Hwang SJ, Liu Y, Sjogren M, van der Pals J, Kalsch H, Muhleisen TW, Nothen MM, Cupples LA, Caslake M, Di Angelantonio E, Danesh J, Rotter JI, Sigurdsson S, Wong Q, Erbel R, Kathiresan S, Melander O, Gudnason V, O'Donnell CJ, Post WS; CHARGE Extracoronary Calcium Working Group. Genetic associations with valvular calcification and aortic stenosis. N Engl J Med. 2013 Feb 7;368(6):503-12. doi: 10.1056/NEJMoa1109034. PMID 23388002